CLINICAL TRIAL: NCT04319978
Title: The Effect of IM Dexamethasone Administered Pre-operatively Versus Post-operatively on Pain and Edema Following Surgical Extraction of Mesio-angularly Impacted Mandibular 3 rd Molars
Brief Title: Dexamethasone Effect on Pain and Edema Following Mandibular 3rd Molar Surgery; Pre-operatively vs Post-operatively
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Arfa baig, Senior Registrar, Dow University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 92 (308) 4448862
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Calcium Dobesilate; Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: A total of 100 patients will be considered in this study which will be equally divided into two groups; group A and group B (50 in each group).Group A will receive dexamethasone 1 hour pre-operatively while group B will receive the same post-operatively.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Group A will receive single dose of dexamethasone IM 8mg 1 hour pre-operatively.
  Interventions: Drug: Dexamethasone injection
- Group B (Active Comparator): Group B will receive a single dose of dexamethasone IM 8mg immediately after surgery.
  Interventions: Drug: Dexamethasone injection

INTERVENTIONS:
Drug: Dexamethasone injection — Dexamethasone is a synthetic corticosteroid. Dexamethasone is an adequate measure for reducing pain and edema in the post-operative recuperation period following 3rd molar surgery. A single dose of IM 8mg dexamethasone will be used for each patient.
  Other Names: Dexa

SUMMARY:
TThis is a comparative clinical study which will be conducted in OMFS department of DIKIOHS, DUHS Ojha Karachi. In this study the investigators will be comparing the effect of dexamethasone on pain and edema when administered pre-operatively vs post-operatively following surgery of impacted lower 3rd molars. Time duration of this study will be 2 months. A total of 100 patients will be considered in this study which will be equally divided into two groups; group A and group B (50 in each group).Group A will receive dexamethasone 1 hour pre-operatively while group B will receive the same post-operatively. All surgeries will be performed by the same maxillofacial surgeon and duration of surgery will be around 30-45 mins.

DETAILED DESCRIPTION:
To compare the effect of dexamethasone (IM; 8mg) administered pre-operatively versus post-operatively on pain and edema following surgical extraction of mesio-angularly impacted mandibular 3rd molars.

This is a comparative clinical study. This study will be conducted in Oral Maxillofacial Surgery department of DIKIOHS, DUHS Teaching Hospital, Ojha, Karachi, Pakistan. Time duration of this study will be 2 months. A total of 100 patients will be considered in the study (50 in each group). Sample size was calculated through OpenEpi, taking mean values of post-operative 3rd day swelling (cm) of group A (12.15±0.78), group B (13.85±0.78) [Ref #], 95% confidence interval (two sided) and 80% of the power of the test. The sample size came out to be 8 patients (4 in each group). The sampling technique is Convenience Sampling. Patients will be randomly distributed into two groups; Group A & Group B. Group A will receive dexamethasone 8mg Intra-muscularly 1 hour pre-operatively while Group B will receive the same immediately after surgery. All surgeries will be performed by the same maxillofacial surgeon and duration of surgery will be around 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming to dental OPD of DIKIOHS, DUHS, Ojha with Mesioangular impactions
* Age of patients: 20-50 years

Exclusion Criteria:

* Patients with known co-morbidities
* Patients allergic to dexamethasone
* Patients with history of recent anti-inflammatory drug intake(NSAIDs, steroids, or antihistamines)
* Pregnant/lactating females

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Change in Edema of face in the mandibular region | Change in edema will be assessed from baseline at 1st, 3rd and 7th day post-operatively
  edema will be assessed using a measuring tape in three facial planes (M1,M2,M3) M1: Tragus of Ear to Corner of Mouth M2: Tragus of Ear to Pogonion M3: Lateral Canthus of Eye to Angle of Mandible.

SECONDARY OUTCOMES:
Change in Intensity of Pain in the extracted site: Visual Analog Scale (VAS) | Change in the intensity of pain will be assessed from baseline to 1st, 3rd and 7th day post-operatively.
  Pain will be assessed using Visual Analog Scale (VAS). VAS is a psychometric response scale which can be used as a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. It is graded from 0 to 10; 0 indicating "No pain" while 10 indicating "excruciating/ unbearable pain"

CONTACTS AND LOCATIONS:
Overall Officials: Arfa Baig, FCPS, Principal Investigator — DIKIOHS, DUHS
Locations (1):
- Dr. Ishrat ul Ebad Khan Institute Of Health Sciences, DUHS, Ojha, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No